CLINICAL TRIAL: NCT06461130
Title: Acute Effect of Dual-task Aerobic Exercise on Cognitive Load and Myocardial Oxygen Consumption in Healthy Sedentary Individuals
Brief Title: Effects of Dual-task Aerobic Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: University of Yalova (Other); Istanbul Gedik University (Other)
Responsible Party: Principal Investigator, ebrar atak, Asst. Prof., University of Yalova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DualTaskwithAerobicTraining
Record Dates: First submitted 2024-06-07; First posted 2024-06-14 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Sedentary Behavior
Keywords: dual task; aerobic training; cardiovascular; cognition
MeSH Terms: conditions — Sedentary Behavior | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double leg dual duty aerobic exercise group (Experimental): During double-leg cycling training, people were made to do dual tasks. Dual-task: aerobic training on a bicycle ergometer + serial sevens In the dual-task condition, participants completed the exercise while simultaneously performing a series of sevens cognitive tasks. Specifically, participants were instructed to serially subtract sevens from a prescribed three-digit number (range 100-300) and read the calculations aloud while performing aerobic exercise.
  Interventions: Other: Study Group
- Double leg standard aerobic exercise group (Active Comparator): In double leg cycling training, both legs; Exercise was performed on the bicycle ergometer, starting with a 5-minute warm-up (25% labor force) on the ergometer before the application, lasting a total of 20 minutes, and continuously training at 70% intensity. Finished with 5 minutes of cooling. Individuals were allowed to maintain a pedaling frequency of 50 rpm, set externally with a metronome.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Study Group — Group of people doing dual tasks during double-leg cycling training.
  Arms: Double leg dual duty aerobic exercise group
Other: Control Group — The group that received only aerobic exercise.
  Arms: Double leg standard aerobic exercise group

SUMMARY:
The aim of this study was to examine the acute effect of dual-task aerobic exercise on cognitive load and myocardial oxygen consumption in healthy sedentary individuals. In this study: 1. Does dual-task exercise applied in addition to aerobic training have an acute effect on cognitive load in healthy sedentary individuals? 2. Does dual-task exercise applied in addition to aerobic training in healthy sedentary individuals have an acute effect on myocardial oxygen consumption, which reflects the indirect oxygen consumption of the heart? The questions were answered.

DETAILED DESCRIPTION:
To find answers to the questions of the study, healthy sedentary participants were randomized into two groups by online randomization method. One of the groups was the group that received only double-leg aerobic exercise. The other group was the double-leg aerobic exercise group integrated with dual-task-oriented training. Before and after the interventions, the blood pressure and pulse rate of the participants were measured, their cognitive functions were evaluated with the MOCA Test, their reaction times were evaluated with the Nelson Reaction Test, and the acute effect of the trainings was examined.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* No comorbidities
* Absence of comorbid diseases of the orthopedic, neurological, cardiopulmonary system
* Participants who have not been involved in another clinical trial in the last 1 month

Exclusion Criteria:

* Participants who had hip, pelvis, knee, ankle surgery in the last year
* Sensory loss
* Participants with leg length inequality
* Participants with known balance disorders in the last three months due to vestibular disorders, pregnancy, concussion
* Presence of systemic disease (diabetes, blood pressure, etc.)
* Those using bronchodilator drugs
* Having a neurological disease
* Not being in good psychological condition

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-07-07 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Cognitive load assessment | Time to acute change in measurements 1 hour before the application and 1 hour after the application.
  Cognitive load change was assessed with the Montreal Cognitive Function Assessment Scale (MOCA).
Myocardial oxygen consumption assessment | Time to acute change in measurements 1 hour before the application and 1 hour after the application.
  Myocardial oxygen consumption was calculated using the Double Product formula of the data obtained from blood pressure and pulse measurement.

SECONDARY OUTCOMES:
Reaction time evaluation | Time to acute change in measurements 1 hour before the application and 1 hour after the application.
  Reaction time was determined by measuring the distance the ruler caught after the ruler was released.

CONTACTS AND LOCATIONS:
Locations (1):
- Ebrar Atak, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided